CLINICAL TRIAL: NCT02080013
Title: Prospective, Randomized Study of Endovenous Segmental Radiofrequency Versus 1320 nm Laser Ablation for the Treatment of Great Saphenous Vein Reflux (RVLAb Study)
Brief Title: Endovenous Radiofrequency Versus Laser Ablation for the Treatment of Great Saphenous Vein Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hossam M. Saleh, A. Prof vascular surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JVS-D-14-00218
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ClosureFast group (Sham Comparator): Radiofrequency Ablation for the Treatment of Great Saphenous Vein Reflux
  Interventions: Other: radiofrequency
- group 1 (Sham Comparator): EVL group Endovenous Laser Ablation for the Treatment of Great Saphenous Vein Reflux
  Interventions: Other: radiofrequency

INTERVENTIONS:
Other: radiofrequency — ClosureFAST
  Other Names: ClosureFAST

SUMMARY:
our aim is to compare early outcomes following EVL 1320 nm and segmental RF in a randomized study.

DETAILED DESCRIPTION:
Endovenous Radiofrequency versus Laser Ablation for the Treatment of Great Saphenous Vein Reflux

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 60 years with incompetent GSVs documented on duplex ultrasound (US; B-mode and color Doppler imaging) were eligible

Exclusion Criteria:

* Exclusion criteria consisted of:
* Current deep vein thrombosis (DVT)
* Thrombus in the vein of interest
* Previous GSV treatment
* Pregnancy
* Known malignancy
* Significant arterial disease (ankle : brachial pressure index below 0•8)
* Use of anticoagulant medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Hossam M. Saleh, PhD, Principal Investigator — Vascular Surgery Department, Ain Shams University